CLINICAL TRIAL: NCT00871572
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Study of LY2409021 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study for Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11095; I1R-MC-GLBE (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Results first posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — adomeglivant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- LY2409021 10 milligrams (mg) (Experimental)
  Interventions: Drug: LY2409021
- LY2409021 30 mg (Experimental)
  Interventions: Drug: LY2409021
- LY2409021 60 mg (Experimental)
  Interventions: Drug: LY2409021

INTERVENTIONS:
Drug: LY2409021 — 4 capsules by mouth taken once daily for 12 weeks
  Arms: LY2409021 10 milligrams (mg); LY2409021 30 mg; LY2409021 60 mg
Drug: Placebo — 4 capsules by mouth once daily for 12 weeks
  Arms: Placebo

SUMMARY:
This drug is being evaluated for possible treatment of type 2 diabetes mellitus. Participation in this study is expected to last up to 18 weeks. A goal of this study is to determine the safety and effectiveness of LY2409021.

ELIGIBILITY:
Inclusion:

* Participants must either be male or a female who cannot become pregnant, who has type 2 diabetes and is either controlling your diabetes through diet and exercise alone, or with diet and exercise taking metformin.
* If participants are male, participants are willing to talk to the study doctor about birth control options during the study and for 3 months after the last dose of study medication.
* Participants must have an Hemoglobin A1c (HbA1c) test of 6.5% to 10%
* Participants must have a body mass index (BMI) between 25 to 40 kilograms/square meter (kg/m²).
* Participants must be willing and able to test your blood sugar levels at home with a blood sugar meter.
* Participants must complete a study diary as instructed by your study doctor and staff and return the study diary as instructed by the study doctor.
* Participants must maintain consistent dietary, physical activity, and sleeping patterns throughout the study.

Exclusion Criteria:

* Insulin, exenatide, or any diabetic medication other than metformin 3 months prior to screening to control you diabetes,
* Medications to increase movement in your digestive tract or that slow movement in your digestive tract
* Over-the-counter drugs or drugs prescribed by your doctor that cause weight loss or high or low blood sugar,
* Chronically use oral glucocorticoids therapy or have received this type of medication within 8 weeks prior to beginning this study,
* Class II and III antiarrhythmic agents (commonly used to prevent or relieve an irregular heartbeat),
* Drugs that damage the liver
* Fibrates and niacin (both commonly used to treat high cholesterol) more than 1 gram/day (gm/day),
* Central nervous stimulants, alcohol intake for males that is more than 2 units per day and for females that is more than 1 unit per day [1 unit=12 ounces (oz) or 360 milliliter (mL) of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits].
* You have had one (1) or more cases of uncontrolled diabetes (very high blood sugars) which required hospitalization in the 6 months prior to the screening visit or have a diagnosis of hypoglycemia (low blood sugar) unawareness.
* You had two (2) or more emergency room visits or were hospitalized for poor control of your diabetes (for example, keto-acidotic episode) in the last 6 months.
* Participants have a problem with your stomach such that it empties slowly (diabetic gastroparesis) or you have had gastric bypass (bariatric) surgery.
* Participants have a personal or family history of pancreatic neoplasia.
* Participants have abnormal lipids (for example triglycerides).
* Participants have had problems with your heart in the past 6 months, such as a heart attack, chest pain (angina), heart failure, heart bypass operation, angioplasty (a medical procedure to open a narrow or clogged blood vessel of the heart) or stent insertion (a procedure to insert a wire mesh tube to prop open a blood vessel after angioplasty), a heart rhythm problem, or a stroke.
* Participants have an elevated or uncontrolled blood pressure.
* Participant's electrocardiogram (ECG, a test that measures the electrical activity of your heart) is outside the normal limits, as determined by the study doctor.
* Participants have a problem with your kidneys or are on dialysis.
* Participants have a problem with your pancreas.
* Participants must not have nor had liver disease (for example, Hepatitis B or C).
* Participants have cancer, except for skin cancer or have been in remission (the absence of disease activity) from cancer for less than 5 years.
* Participants have a serious or uncontrolled health problems (other than type 2 diabetes), blood disorders or laboratory tests that in the opinion of the doctor, could interfere with understanding the results of this study. The doctor will let you know if this applies to you.
* Participants previously completed or withdrew from this study or any other study investigating LY2409021.
* Participants are allergic to the study drug or other related drugs. You cannot be in this study if you are a woman and you possibly could become pregnant during this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (19):
- United States (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buena Park, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntington Park, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westlake Village, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jupiter, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Port Richey, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madisonville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rapid City, South Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norfolk, Virginia
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aschaffenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saarlouis
- Lithuania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaunas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vilnius

REFERENCES:
- [Derived] Kazda CM, Ding Y, Kelly RP, Garhyan P, Shi C, Lim CN, Fu H, Watson DE, Lewin AJ, Landschulz WH, Deeg MA, Moller DE, Hardy TA. Evaluation of Efficacy and Safety of the Glucagon Receptor Antagonist LY2409021 in Patients With Type 2 Diabetes: 12- and 24-Week Phase 2 Studies. Diabetes Care. 2016 Jul;39(7):1241-9. doi: 10.2337/dc15-1643. Epub 2015 Dec 17. PMID 26681715

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo was administered orally once daily as 4 capsules for 12 weeks.
- 10 mg LY2409021: 10 milligram (mg) LY2409021 was administered orally once daily as 4 capsules of 2.5 mg LY2409021 for 12 weeks.
- 30 mg LY2409021: 30 mg LY2409021 was administered orally once daily as 2 capsules of 15 mg LY2409021 and 2 capsules of placebo for 12 weeks.
- 60 mg LY2409021: 60 mg LY2409021 was administered orally once daily as 4 capsules of 15 mg LY2409021 for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Started | 10 | 17 | 34 | 26
≥1 Post Baseline Value by Assigned Group | 9 | 17 | 34 | 25
Received at Least 1 Dose of Study Drug | 9 | 17 | 34 | 25
Completed | 8 | 11 | 30 | 19
Not Completed | 2 | 6 | 4 | 7
Not completed — Adverse Event | 0 | 2 | 0 | 3
Not completed — Investigator Decision | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Sponsor Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 10 mg LY2409021: 10 mg LY2409021 was administered orally once daily as 4 capsules of 2.5 mg LY2409021 for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021 | Total
Number analyzed (Participants) | 10 | 17 | 34 | 26 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (4.92) | 53.3 (10.20) | 52.0 (10.88) | 52.5 (6.41) | 52.3 (8.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 18 | 18 | 47
  Male | 5 | 11 | 16 | 8 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 10 | 15 | 16 | 48
  Not Hispanic or Latino | 3 | 7 | 19 | 10 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 9 | 9 | 23
  Asian | 0 | 2 | 1 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 5 | 3 | 15
  White | 5 | 7 | 18 | 11 | 41
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 17 | 34 | 26 | 87

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Glycosylated Hemoglobin A1c (HbA1c)
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was calculated using a mixed-model repeated measures analysis (MMRM) that included terms for treatment group, baseline HbA1c, metformin use, visit, and visit-by-treatment interaction.
Time Frame: Baseline, Week 12
Population: Modified Intent-to-Treat (mITT): All randomized participants with at least 1 post baseline HbA1c measurement and analyzed according to the assigned treatment.
Measure: Least Squares Mean (90% Confidence Interval); unit: percentage of HbA1c
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Number analyzed (Participants) | 8 | 11 | 31 | 19
percentage of HbA1c | 0.11 [-0.44 to 0.65] | -0.83 [-1.28 to -0.38] | -0.65 [-0.93 to -0.37] | -0.66 [-1.00 to -0.31]
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.0296, Mixed Models Analysis; Mean Difference (Final Values) = -0.94, 90% CI 2-sided [-1.64 to -0.23]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.0418, Mixed Models Analysis; Mean Difference (Final Values) = -0.76, 90% CI 2-sided [-1.37 to -0.15]
Statistical Analysis 3: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.0514, Mixed Models Analysis; Mean Difference (Final Values) = -0.76, 90% CI 2-sided [-1.41 to -0.12]

2. Secondary Outcome: Change From Baseline Values for Fasting Blood Glucose (FBG)
Description: LS mean was calculated using a MMRM that included terms for treatment group, baseline value, metformin use, visit, and visit-by-treatment interaction.
Time Frame: Baseline, Week 12
Population: mITT: All randomized participants with at least 1 post baseline FBG measurement and analyzed according to the assigned treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimoles/liter (mmol/L)
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Number analyzed (Participants) | 8 | 10 | 31 | 20
millimoles/liter (mmol/L) | 1.19 [-0.93 to 3.32] | -0.43 [-2.30 to 1.44] | -0.67 [-1.76 to 0.42] | -1.22 [-2.55 to 0.11]
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.2565, Mixed Models Analysis; Mean Difference (Final Values) = -1.62, 95% CI 2-sided [-4.46 to 1.21]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.1245, Mixed Models Analysis; Mean Difference (Final Values) = -1.86, 95% CI 2-sided [-4.25 to 0.53]
Statistical Analysis 3: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.0594, Mixed Models Analysis; Mean Difference (Final Values) = -2.41, 95% CI 2-sided [-4.92 to 0.10]

3. Secondary Outcome: Change From Baseline for Glucose Area Under the Curve (AUC) From Oral Glucose Tolerance Test (OGTT)
Description: LS mean was calculated using analysis of covariance (ANCOVA) model that included terms for treatment group, baseline value and metformin use.
Time Frame: Baseline, Week 12
Population: mITT: All randomized participants with at least 1 post baseline OGTT measurement and analyzed according to the assigned treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Number analyzed (Participants) | 6 | 10 | 29 | 19
mmol/L | 172.89 [-117.67 to 463.46] | 48.34 [-178.20 to 274.88] | -165.74 [-297.35 to -34.14] | -293.94 [-458.59 to -129.29]
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.4978, ANCOVA; Mean Difference (Final Values) = -124.56, 95% CI 2-sided [-490.02 to 240.90]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.0372, ANCOVA; Mean Difference (Final Values) = -338.64, 95% CI 2-sided [-656.55 to -20.72]
Statistical Analysis 3: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.0068, ANCOVA; Mean Difference (Final Values) = -466.83, 95% CI 2-sided [-799.48 to -134.18]

4. Secondary Outcome: Change From Baseline to Endpoint for Fasting Triglycerides
Description: LS mean was calculated using ANCOVA model that included terms for treatment group, baseline value and metformin use.
Time Frame: Baseline, Week 12
Population: mITT: All randomized participants with at least 1 post baseline fasting triglyceride measurement and analyzed according to the assigned treatment.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Number analyzed (Participants) | 7 | 10 | 30 | 19
mmol/L | 0.1 (0.24) | 0.2 (0.20) | 0.2 (0.12) | 0 (0.14)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.814, ANCOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.5 to 0.7]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.681, ANCOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.4 to 0.7]
Statistical Analysis 3: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.715, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.7 to 0.5]

5. Secondary Outcome: Total and Sub-Domain Scores of Diabetes Symptom Checklist-Revised (DSC-R)
Description: The DSC-R was a participant completed questionnaire that was designed to assess the presence and perceived burden of diabetes-related symptoms. Participants were asked to recall the last 4 weeks and consider each symptom/item in terms of whether they experienced it and if so, how troublesomeness it was. Participants were to consider troublesomeness of the symptom on a 1 (not at all) to 5 (extremely) point scale. There were a total of 34 items, grouped into 8 subscales: cardiovascular (4 items), psychological-cognitive distress (4 items), psychological-fatigue (4 items), hyperglycemic (4 items), hypoglycemic (3 items), neurological-pain (4 items), neurological-sensory (6 items) and visual (5 items). Sub-domain score calculated as: (sum of item scores) divided by (number of items), scores ranged from 1 to 5. Total score was the sum of all sub-domains and ranged from 8 to 40. Higher scores of total and subscales indicated worsened symptoms.
Time Frame: Baseline, Week 12
Population: mITT: All randomized participants with at least 1 post baseline DSC-R measurement and analyzed according to the assigned treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Number analyzed (Participants) | 10 | 17 | 34 | 36
units on a scale
  Cardiovascular: number analyzed (Participants) | 1 | 4 | 4 | 5
  Cardiovascular | 2.5 (NA) — One (1) participant analyzed, therefore, the standard deviation (SD) was not calculated. | 1.52 (0.372) | 1.52 (0.475) | 1.69 (0.586)
  Hyperglycemic: number analyzed (Participants) | 2 | 5 | 16 | 10
  Hyperglycemic | 3.18 (1.517) | 2.79 (1.086) | 2.30 (0.437) | 2.37 (0.563)
  Hypoglycemic: number analyzed (Participants) | 2 | 4 | 9 | 4
  Hypoglycemic | 1.50 (0707) | 2.42 (1.258) | 2.50 (0.980) | 2.00 (1.277)
  Neurological-Pain: number analyzed (Participants) | 1 | 4 | 8 | 6
  Neurological-Pain | 2.00 (NA) — One (1) participant analyzed, therefore, the SD was not calculated. | 1.91 (0.717) | 1.88 (0.396) | 1.80 (0636)
  Neurological-Sensory: number analyzed (Participants) | 3 | 5 | 7 | 7
  Neurological-Sensory | 2.39 (0.438) | 1.89 (0.587) | 2.35 (0.596) | 2.11 (0.893)
  Visual: number analyzed (Participants) | 1 | 4 | 7 | 5
  Visual | 1.00 (NA) — One (1) participant analyzed, therefore, the SD was not calculated. | 2.45 (1.172) | 2.03 (0.812) | 2.05 (1.160)
  Psychological-Cognitive: number analyzed (Participants) | 2 | 4 | 7 | 5
  Psychological-Cognitive | 1.61 (0.860) | 2.31 (0.875) | 2.37 (0.967) | 1.69 (0.636)
  Psychological-Fatigue: number analyzed (Participants) | 2 | 7 | 15 | 8
  Psychological-Fatigue | 1.91 (0.219) | 2.06 (0.734) | 2.33 (0.584) | 2.07 (0.500)
  Total | NA (NA) — Total was not calculated due to too much missing subdomain data as per the protocol. | NA (NA) — Total was not calculated due to too much missing subdomain data as per the protocol. | NA (NA) — Total was not calculated due to too much missing subdomain data as per the protocol. | NA (NA) — Total was not calculated due to too much missing subdomain data as per the protocol.

6. Secondary Outcome: Change From Baseline in the Diabetes Medicines Survey Perceived Effectiveness and Physical Side-Effects (Differences Between Perceptions About Medication-Diabetes Scores Between Placebo and LY2409021)
Description: The Diabetes Medicines Survey was a participant reported questionnaire consisting of 25 items: perceived effectiveness of diabetes medicines (items 1-10) and physical side-effects (items 11-25). Both domains had a scores range from 1 (all of the time) to 4 (none of the time) and a possible total scores range from 25 to 100. Lower scores for perceived effectiveness items indicated a better perceived effectiveness. Lower scores for physical side-effects items indicated a greater frequency of physical side-effects.
Time Frame: Baseline, Week 12
Population: mITT: All randomized participants with at least 1 post baseline Diabetes Medicines Survey measurement and analyzed according to the assigned treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Number analyzed (Participants) | 8 | 11 | 30 | 19
units on a scale
  Medication controlling blood sugar(BS) | 1.75 (0.886) | 2.00 (0.894) | 1.77 (0.679) | 1.53 (0.697)
  Meeting medical needs | 1.75 (0.886) | 2.09 (0.831) | 1.80 (0.805) | 1.58 (0.769)
  Medication working well | 1.75 (0.886) | 2.00 (0.894) | 1.70 (0.794) | 1.63 (0.831)
  Medication giving good results | 1.88 (0.835) | 2.00 (0.894) | 1.87 (0.776) | 1.58 (0692)
  Medication making me feel better | 2.00 (1.069) | 2.09 (0.831) | 1.90 (0.712) | 1.84 (0.688)
  Medication taking care of illness | 2.00 (1.069) | 2.09 (0.831) | 1.83 (0.834) | 1.58 (0.692)
  Medication therapy is failing: number analyzed (Participants) | 8 | 11 | 29 | 19
  Medication therapy is failing | 3.63 (0.744) | 3.18 (0.874) | 3.17 (0.928) | 3.58 (0769)
  Medication giving 24-hour control: number analyzed (Participants) | 8 | 11 | 29 | 19
  Medication giving 24-hour control | 2.13 (1.126) | 2.27 (1.104) | 2.03 (0.823) | 1.68 (0.671)
  Medication therapy is effective | 1.88 (0.835) | 2.09 (0.944) | 1.87 (0.730) | 1.74 (0.733)
  Medication keeping BS stable | 2.00 (0.926) | 2.18 (0.982) | 1.97 (0.718) | 1.68 (0.671)
  Side Effect: Constipation | 3.88 (0.354) | 3.18 (1.168) | 3.83 (0.379) | 3.63 (0.761)
  Side Effect: Feet or hands swelling | 3.75 (0.463) | 3.91 (0.302) | 3.80 (0.407) | 3.84 (0.375)
  Side Effect: Headaches | 3.63 (0.518) | 3.45 (0.688) | 3.60 (0563) | 3.79 (0.419)
  Side Effect: Weight gain | 3.63 (0.518) | 3.73 (0.467) | 3.57 (0.728) | 3.79 (0.419)
  Side Effect: Dizziness/Lightheaded | 3.75 (0.463) | 3.73 (0.467) | 3.90 (0.403) | 3.89 (0.315)
  Side Effect: Muscle Cramps | 3.88 (0.354) | 3.64 (0.809) | 3.87 (0.346) | 3.58 (0.769)
  Side Effect: Bloating | 3.63 (0.518) | 3.82 (0.405) | 3.83 (0.379) | 3.79 (0.419)
  Side Effect: Diarrhea | 3.38 (0.744) | 3.73 (0.467) | 3.70 (0.596) | 3.74 (0.452)
  Side Effect: Heartburn: number analyzed (Participants) | 8 | 11 | 29 | 19
  Side Effect: Heartburn | 3.75 (0.463) | 3.73 (0.647) | 3.72 (0.528) | 3.79 (0.535)
  Side Effect: Excessive Sweating | 3.75 (0.463) | 3.64 (0.809) | 3.77 (0.568) | 3.79 (0.535)
  Side Effect: Itching | 3.88 (0.354) | 3.73 (0.467) | 3.90 (0.403) | 3.84 (0.501)
  Side Effect: Hypoglycemia | 4.00 (0.000) | 3.82 (0.405) | 3.90 (0.305) | 3.89 (0.315)
  Side Effect: Stomach Pain | 3.75 (0.707) | 3.73 (0.647) | 3.93 (0.254) | 3.84 (0.375)
  Side Effect: Upset Stomach | 3.63 (0.744) | 4.00 (0.000) | 3.90 (0.305) | 3.79 (0.535)
  Side Effect: Muscle Soreness | 3.75 (0.463) | 3.82 (0.603) | 3.77 (0.504) | 3.63 (0.597)

7. Secondary Outcome: Change From Baseline Values for 7-Point Self-Monitored Blood Glucose (SMBG) Profiles
Description: Participants obtained 7-point SMBG values immediately before and 2 hours after each meal and at bedtime. LS mean was calculated using a MMRM that included terms for treatment group, baseline value, metformin use, visit, and visit-by-treatment interaction.
Time Frame: Baseline, Week 12
Population: mITT: All randomized participants with at least 1 post baseline 7-Point SMBG measurement and analyzed according to the assigned treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams/deciliter (mg/dL)
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Number analyzed (Participants) | 8 | 11 | 28 | 18
milligrams/deciliter (mg/dL)
  Pre-Morning Meal Fasting | 13.46 [-2.23 to 29.15] | -10.09 [-23.27 to 3.08] | -21.82 [-30.19 to -13.44] | -25.86 [-36.20 to -15.52]
  2 Hours After Morning Meal | -27.48 [-49.06 to -5.90] | -33.90 [-52.13 to -15.67] | -35.68 [-46.98 to -24.38] | -34.68 [-48.61 to -20.75]
  Pre Mid-Day Meal | 16.43 [-2.08 to 34.94] | -19.39 [-35.07 to -3.71] | -16.72 [-26.55 to -6.90] | -21.44 [-33.55 to -9.33]
  2 Hours After Mid-Day Meal | -6.86 [-27.59 to 13.88] | -35.34 [-52.73 to -17.94] | -22.51 [-33.57 to -11.46] | -29.42 [-42.91 to -15.92]
  Pre Evening Meal | 28.16 [5.23 to 51.08] | -16.62 [-36.01 to 2.77] | -26.29 [-38.48 to -14.11] | -18.03 [-33.00 to -3.07]
  2 Hours After Evening Meal | 12.02 [-11.55 to 35.58] | -27.80 [-47.30 to -8.31] | -31.78 [-44.13 to -19.42] | -27.54 [-42.73 to -12.34]
  Bedtime | 17.19 [-5.34 to 39.72] | -19.69 [-38.75 to -0.63] | -29.31 [-41.14 to -17.48] | -24.88 [-39.84 to -9.92]
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.0248, Mixed Models Analysis — P-value is for Pre-Morning Meal (fasting); Mean Difference (Final Values) = -23.56, 95% CI 2-sided [-44.03 to -3.09]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — P-value is for Pre-Morning Meal (fasting); Mean Difference (Final Values) = -35.28, 95% CI 2-sided [-53.08 to -17.48]
Statistical Analysis 3: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value is for Pre-Morning Meal (fasting); Mean Difference (Final Values) = -39.32, 95% CI 2-sided [-58.12 to -20.53]
Statistical Analysis 4: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.6513, Mixed Models Analysis — P-value is for 2 Hours After Morning Meal; Mean Difference (Final Values) = -6.42, 95% CI 2-sided [-34.66 to 21.82]
Statistical Analysis 5: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.5045, Mixed Models Analysis — P-value is for 2 Hours After Morning Meal; Mean Difference (Final Values) = -8.20, 95% CI 2-sided [-32.61 to 16.21]
Statistical Analysis 6: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.5774, Mixed Models Analysis — P-value is for 2 Hours After Morning Meal; Mean Difference (Final Values) = -7.20, 95% CI 2-sided [-32.90 to 18.49]
Statistical Analysis 7: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.0045, Mixed Models Analysis — P-value is for Pre-Mid-Day Meal; Mean Difference (Final Values) = -35.81, 95% CI 2-sided [-60.10 to -11.53]
Statistical Analysis 8: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.0024, Mixed Models Analysis — P-value is for Pre-Mid-Day Meal; Mean Difference (Final Values) = -33.15, 95% CI 2-sided [-54.10 to -12.21]
Statistical Analysis 9: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis — P-value is for Pre-Mid-Day Meal; Mean Difference (Final Values) = -37.87, 95% CI 2-sided [-59.98 to -15.75]
Statistical Analysis 10: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.0389, Mixed Models Analysis — P-value is for 2 Hours After Mid-Day Meal; Mean Difference (Final Values) = -28.48, 95% CI 2-sided [-55.47 to -1.49]
Statistical Analysis 11: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.1896, Mixed Models Analysis — P-value is for 2 Hours After Mid-Day Meal; Mean Difference (Final Values) = -15.65, 95% CI 2-sided [-39.24 to 7.94]
Statistical Analysis 12: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.0729, Mixed Models Analysis — P-value is for 2 Hours After Mid-Day Meal; Mean Difference (Final Values) = -22.56, 95% CI 2-sided [-47.28 to 2.16]
Statistical Analysis 13: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.0041, Mixed Models Analysis — P-value is for Pre Evening Meal; Mean Difference (Final Values) = -44.78, 95% CI 2-sided [-74.79 to -14.77]
Statistical Analysis 14: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value is for Pre Evening Meal; Mean Difference (Final Values) = -54.45, 95% CI 2-sided [-80.42 to -28.48]
Statistical Analysis 15: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis — P-value is for Pre Evening Meal; Mean Difference (Final Values) = -46.19, 95% CI 2-sided [-73.57 to -18.81]
Statistical Analysis 16: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.0118, Mixed Models Analysis — P-value is for 2 Hours After Evening Meal; Mean Difference (Final Values) = -39.82, 95% CI 2-sided [-70.51 to -9.13]
Statistical Analysis 17: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis — P-value is for 2 Hours After Evening Meal; Mean Difference (Final Values) = -43.80, 95% CI 2-sided [-70.42 to -17.18]
Statistical Analysis 18: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.0065, Mixed Models Analysis — P-value is for 2 Hours After Evening Meal; Mean Difference (Final Values) = -39.56, 95% CI 2-sided [-67.63 to -11.48]
Statistical Analysis 19: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.0154, Mixed Models Analysis — P-value is for Bedtime; Mean Difference (Final Values) = -36.88, 95% CI 2-sided [-66.43 to -7.33]
Statistical Analysis 20: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis — P-value is for Bedtime; Mean Difference (Final Values) = -46.50, 95% CI 2-sided [-71.93 to -21.07]
Statistical Analysis 21: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.0029, Mixed Models Analysis — P-value is for Bedtime; Mean Difference (Final Values) = -42.07, 95% CI 2-sided [-69.13 to -15.01]

8. Secondary Outcome: Change From Baseline Values for Fasting Insulin
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: mITT: All randomized participants with at least 1 post baseline fasting insulin measurement and analyzed according to the assigned treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: picomole/liter (pmol/L)
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Number analyzed (Participants) | 7 | 11 | 30 | 19
picomole/liter (pmol/L) | -10.91 [-56.58 to 34.76] | 14.71 [-21.17 to 50.59] | -5.51 [-27.50 to 16.49] | 13.34 [-14.08 to 40.76]
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.3815, Mixed Models Analysis; Mean Difference (Final Values) = 25.62, 95% CI 2-sided [-32.44 to 83.68]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.8315, Mixed Models Analysis; Mean Difference (Final Values) = 5.40, 95% CI 2-sided [-45.12 to 55.93]
Statistical Analysis 3: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.3658, Mixed Models Analysis; Mean Difference (Final Values) = 24.25, 95% CI 2-sided [-28.93 to 77.44]

9. Secondary Outcome: Change From Baseline Values for Fasting Glucagon
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: mITT: All randomized participants with at least 1 post baseline fasting glucagon measurement and analyzed according to the assigned treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Number analyzed (Participants) | 8 | 11 | 31 | 19
pmol/L | -2.36 [-70.57 to 65.85] | 52.71 [-1.84 to 107.25] | 87.32 [52.35 to 122.30] | 104.90 [61.28 to 148.52]
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.2131, Mixed Models Analysis; Mean Difference (Final Values) = 55.06, 95% CI 2-sided [-32.24 to 142.37]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.0220, Mixed Models Analysis; Mean Difference (Final Values) = 89.68, 95% CI 2-sided [13.27 to 166.10]
Statistical Analysis 3: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.0101, Mixed Models Analysis; Mean Difference (Final Values) = 107.26, 95% CI 2-sided [26.29 to 188.22]

10. Secondary Outcome: Change From Baseline Values for Fasting Glucagon-Like Peptide 1 (GLP-1)
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: mITT: All randomized participants with at least 1 post baseline fasting GLP-1 measurement and analyzed according to the assigned treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Number analyzed (Participants) | 8 | 11 | 29 | 19
pmol/L | -1.43 [-3.44 to 0.58] | 0.44 [-1.24 to 2.13] | 0.61 [-0.45 to 1.66] | 0.28 [-1.00 to 1.57]
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.1596, Mixed Models Analysis; Mean Difference (Final Values) = 1.87, 95% CI 2-sided [-0.75 to 4.49]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.0791, Mixed Models Analysis; Mean Difference (Final Values) = 2.03, 95% CI 2-sided [-0.24 to 4.31]
Statistical Analysis 3: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.1564, Mixed Models Analysis; Mean Difference (Final Values) = 1.71, 95% CI 2-sided [-0.67 to 4.10]

11. Secondary Outcome: Change From Baseline for Insulin AUC From OGTT
Description: LS mean was calculated using an ANCOVA that included terms for treatment group, baseline value and metformin use.
Time Frame: Baseline, Week 12
Population: mITT: All randomized participants with at least 1 post baseline AUC from OGTT measurement and analyzed according to the assigned treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Number analyzed (Participants) | 6 | 10 | 28 | 17
pmol/L | 2357.88 [-14350.13 to 19065.88] | 10376.38 [-2525.67 to 23278.44] | 7532.72 [-199.74 to 15265.19] | 20511.79 [10583.81 to 30439.77]
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.4500, ANCOVA; Mean Difference (Final Values) = 8018.51, 95% CI 2-sided [-13104.14 to 29141.16]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.5739, ANCOVA; Mean Difference (Final Values) = 5174.85, 95% CI 2-sided [-13158.65 to 23508.35]
Statistical Analysis 3: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.0653, ANCOVA; Mean Difference (Final Values) = 18153.92, 95% CI 2-sided [-1188.23 to 37496.06]

12. Secondary Outcome: Change From Baseline for C-Peptide AUC From OGTT
Description: LS mean was calculated using an ANCOVA model that included terms for treatment group, baseline value and metformin use.
Time Frame: Baseline, Week 12
Population: mITT: all randomized participants with at least 1 post baseline C-peptide AUC from OGTTmeasurement and analyzed according to the assigned treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Number analyzed (Participants) | 6 | 11 | 29 | 19
pmol/L | 20380.84 [-38421.86 to 79183.54] | 38475.16 [-4765.49 to 81715.81] | 26164.43 [-535.64 to 52864.50] | 56599.82 [23333.38 to 89866.26]
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.6209, ANCOVA; Mean Difference (Final Values) = 18094.32, 95% CI 2-sided [-54734.08 to 90922.71]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.8581, ANCOVA; Mean Difference (Final Values) = 5783.59, 95% CI 2-sided [-58650.71 to 70217.89]
Statistical Analysis 3: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.2850, ANCOVA; Mean Difference (Final Values) = 36218.98, 95% CI 2-sided [-30955.50 to 103393.46]

13. Secondary Outcome: Change From Baseline to Endpoint for Low Density Lipoprotein (LDL)
Description: Fasting LDL LS mean was calculated using ANCOVA that included terms for baseline and treatment.
Time Frame: Baseline, Week 12
Population: mITT: All randomized participants with at least 1 post baseline fasting LDL measurement and analyzed according to the assigned treatment; last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Number analyzed (Participants) | 8 | 16 | 31 | 21
mmol/L | 0.4 (0.21) | 0.3 (0.15) | 0.2 (0.11) | 0.3 (0.13)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.584, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.7 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.426, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.7 to 0.3]
Statistical Analysis 3: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.657, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.6 to 0.4]

14. Secondary Outcome: Change From Baseline to Endpoint for High Density Lipoprotein (HDL)
Description: Fasting HDL LS mean was calculated using ANCOVA that included terms for baseline and treatment.
Time Frame: Baseline, Week 12
Population: mITT: All randomized participants with at least 1 post baseline fasting HDL measurement and analyzed according to the assigned treatment; LOCF.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Number analyzed (Participants) | 8 | 16 | 32 | 22
mmol/L | -0.1 (0.11) | 0 (0.07) | 0.1 (0.05) | 0 (0.06)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.365, ANCOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.1 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.191, ANCOVA; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.1 to 0.4]
Statistical Analysis 3: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.297, ANCOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.1 to 0.4]

15. Secondary Outcome: Change From Baseline to Endpoint for Non-HDL Cholesterol
Description: Fasting non-HDL cholesterol LS mean was calculated using ANCOVA that included terms for baseline and treatment.
Time Frame: Baseline, Week 12
Population: mITT: All randomized participants with at least 1 post baseline fasting non-HDL cholesterol measurement and analyzed according to the assigned treatment; LOCF.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Number analyzed (Participants) | 8 | 16 | 32 | 22
mmol/L | 0.5 (0.24) | 0.3 (0.17) | 0.3 (0.12) | 0.3 (0.14)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.523, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.8 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.476, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.7 to 0.3]
Statistical Analysis 3: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.634, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.7 to 0.4]

16. Secondary Outcome: Change From Baseline to Endpoint for Total Cholesterol
Description: Fasting total cholesterol LS mean was calculated using ANCOVA that included terms for baseline and treatment.
Time Frame: Baseline, Week 12
Population: mITT: All randomized participants with at least 1 post baseline fasting total cholesterol measurement and analyzed according to the assigned treatment; LOCF.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Number analyzed (Participants) | 9 | 16 | 33 | 23
mmol/L | 0.3 (0.24) | 0.3 (0.18) | 0.3 (0.12) | 0.4 (0.15)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY2409021; Test type: Superiority or Other; p = 0.919, ANCOVA; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.6 to 0.6]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY2409021; Test type: Superiority or Other; p = 0.864, ANCOVA; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.5 to 0.6]
Statistical Analysis 3: Comparison: Placebo vs 60 mg LY2409021; Test type: Superiority or Other; p = 0.726, ANCOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.5 to 0.7]

ADVERSE EVENTS:
Arm/Group | Placebo | 10 mg LY2409021 | 30 mg LY2409021 | 60 mg LY2409021
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/17 | 0/34 | 1/25
Other Adverse Events (participants affected / at risk) | 6/9 | 14/17 | 25/34 | 18/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | 10 mg LY2409021 (N=17) | 30 mg LY2409021 (N=34) | 60 mg LY2409021 (N=25)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | 10 mg LY2409021 (N=17) | 30 mg LY2409021 (N=34) | 60 mg LY2409021 (N=25)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (6) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 5 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram t wave abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 2 (3) | 2 (2)
Weight increased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 2 (4) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 2 (4) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (3) | 3 (3)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days